CLINICAL TRIAL: NCT06702683
Title: Study on the Correlation Between Blood Concentration of Sintilimab and Related Predictors with Efficacy and Adverse Reactions in Patients with Advanced Gastric Cancer
Brief Title: The Correlation Between Blood Concentration of Sintilimab and Efficacy and Adverse Reactions in Patients with Advanced Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Lin Liu (Other)
Responsible Party: Sponsor-Investigator, Lin Liu, Chief physician of Oncology Department, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Other Study IDs: 2022ZDSYLL329-P01
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Gastric Carcinoma; Gastric Neoplasm; Gastric (cardia, Body) Cancer; Gastric Cancer Adenocarcinoma Metastatic
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Compared with other anti-tumor drugs, immune checkpoint inhibitors (ICIs) have their own unique pharmacokinetics (PK) and pharmacodynamics (PD), and affect patient clinical outcomes. However, at present, the data on the PK and PD characteristics of ICIs in the Chinese population are still lacking, thus further clinical trials are needed to verify them. At the same time, a large proportion of patients have no response to ICIs or the efficacy is poor, and even bring greater side effects, so it is particularly important to find effective biomarkers to predict the efficacy and adverse reactions of patients with ICIs treatment.The purpose of this study is to explore the correlation between blood concentration of Sintilimab and related predictors with efficacy and adverse reactions in patients with advanced gastric cancer so as to provide clinical reference for individualized treatment of patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

A. Patients who were diagnosed with gastric adenocarcinoma or gastroesophageal junction adenocarcinoma; B. Patients who plan to be treated with Sintilimab; C.ECOG score of 0-2; D. Expected survival ≥3 months; E. The patient who have good compliance, follow-up, and can cooperate with relevant treatment and examination; F. Agree to participate in the study and sign the informed consent

Exclusion Criteria:

A. Patients who clinical information and data are incomplete; B. Patients who treated with immune checkpoint inhibitors within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced gastric cancer patients treated with sindilizumab in the Oncology Department of Zhongda Hospital Affiliated to Southeast University
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
blood concentration of Sintilimab | From February 2023 to June 2025

SECONDARY OUTCOMES:
the cytokines in peripheral blood | From February 2023 to June 2025
  the cytokines in peripheral blood including:IL -1β, IL-2, IL-4, IL-6, IL-8, IL-10, IFN-γ, TNF-α, TNF-β
Inflammatory biomarkers in peripheral blood | From February 2023 to June 2025
  Inflammatory biomarkers in peripheral blood including:NLR, PLR, LMR/MLR, LIPI
T lymphocyte subsets in peripheral blood | From February 2023 to June 2025
  T lymphocyte subsets in peripheral blood including: CD4, CD8, Th1, Th9, Th17
Fatty acid and bile acid metabolism | From February 2023 to June 2025
  Fatty acid and bile acid metabolism:short-chain fatty acid including:ursodeoxycholic acid, short-chain fatty acid, polyunsaturated fatty acids
Anti-drug antibody | From February 2023 to June 2025
  ADA

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No